CLINICAL TRIAL: NCT07219524
Title: Problem-Solving Skills Training for Parents of Children Undergoing Hematopoietic Stem Cell Transplantation: A Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Los Angeles (Other)
Responsible Party: Principal Investigator, Bemis, Heather, Assistant Professor of Clinical Pediatrics, Children's Hospital Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CHLA-20-00276
Record Dates: First submitted 2025-10-20; First posted 2025-10-22 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Stem Cell Transplantation
Keywords: Problem-Solving Skills Training; Parent or caregiver support; behavioral intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Standard of care.
- Problem-Solving Skills Training (Experimental): Bright ideas problem solving skills intervention.
  Interventions: Behavioral: Bright Ideas Problem-Solving Skills Training

INTERVENTIONS:
Behavioral: Bright Ideas Problem-Solving Skills Training — Intervention materials include instructor and user manuals, a brochure, and worksheets to be completed by the parent caregiver, initially with the help of the interventionist, during four weekly face-to-face (F2F) sessions
  Arms: Problem-Solving Skills Training

SUMMARY:
The goal of this clinical trial is to test the feasibility and acceptability of the Bright IDEAS problem-solving skills training (PSST) intervention for parents of children undergoing hematopoietic stem cell transplantation (HSCT). The main question aims to answer:

* Determine the feasibility and acceptability of a multimodal PSST intervention for English and Spanish-speaking parents of children and adolescents undergoing autologous and allogeneic HSCT using a randomized controlled trial design and mixed methods approach to evaluation
* To evaluate the effectiveness of a PSST intervention on PSS acquisition and psychological distress compared to a control group of parents receiving non-directive psychosocial care (n=25).
* To explore the effect of the parent PSST on child quality of life (QoL) and self-reported symptoms, mediated by parent psychological distress

If there is a comparison group: Researchers will compare PSST intervention usual or standard psychosocial care.

Participants will complete 6-8 sessions of intervention. All participants will complete surveys.

ELIGIBILITY:
Children

Inclusion Criteria:

* Male and females of any race or ethnicity, ages 0 to 21 years
* Allogeneic or autologous HSCT planned with reduced intensity or myeloablative conditioning

Exclusion Criteria:

* Concurrent enrollment on a research study testing psychoeducational interventions for parents and/or patients

Parent

Inclusion Criteria:

* One parent or primary caregiver per child
* Able to speak, read, and write English or Spanish, and give informed consent

Exclusion Criteria:

* Child or adolescent refusal to participate
* Parent age less than 18 years.

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2020-11-11 (Actual); Primary Completion 2023-05-23 (Actual); Study Completion 2023-05-23 (Actual)

PRIMARY OUTCOMES:
Feasibility of Bright IDEAS for parents | Baseline to 180 days
  Percent eligible participants who consent/assent to participate and Number of sessions completed by enrolled participants.
Bright IDEAS Acceptability | Between day 60 and day 90
  Qualitative Interviews will assess participant satisfaction with the intervention format, timing, and content; impact; barriers; and suggestions for refinement.

SECONDARY OUTCOMES:
Parent Problem Solving Skills | Baseline to 180 days
  Social Problem-Solving Skills Inventory-Revised Short Form
Parent Negative Affectivity | Baseline to 180 days
  Profile of Mood States Short Form
Parent Anxiety | Baseline to 180 days
  Beck Anxiety Inventory
Parent Depression | Baseline to 180 days
  Beck Depression Inventory
Parent Post-traumatic Stress | Baseline to 180 days
  Impact of events scale revised
Children Symptom Burden | Baseline to 180 days
  Memorial Symptoms Assessment Scale (Child Version & Parent Proxy for children ages 2-6 years)
Children Health-Related Quality of Life | Baseline to 180 days
  PedsQL Cancer Module (Child Version & Parent Proxy for children ages 2-4 years)

CONTACTS AND LOCATIONS:
Overall Officials: Heather Bemis, Principal Investigator — Children's Hospital Los Angeles
Locations (1):
- Children's Hospital Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No